CLINICAL TRIAL: NCT05037344
Title: Internet-based Cognitive Behavioral Psychotherapy for Children and Adolescents With Obsessive-compulsive Disorder II
Brief Title: iCBT for Children and Adolescents With Obsessive-compulsive Disorder II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, PD Dr. Annette Conzelmann, PD Dr. Annette Conzelmann, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AZ 53-5400.1-004/44
Record Dates: First submitted 2021-07-31; First posted 2021-09-08 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Psychotherapy Intervention Evaluation
Keywords: cognitive-behavioral psychotherapy; obsessive-compulsive disorder; internet-based
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-based psychotherapy (Experimental): 16 weeks of internet-based cognitive behavioral therapy
  Interventions: Behavioral: Cognitive-behavioral psychotherapy
- Internet-based psychotherapy waiting group (Active Comparator): 16 weeks of internet-based cognitive bahavioral therapy after waiting of 16 weeks
  Interventions: Behavioral: Cognitive-behavioral psychotherapy

INTERVENTIONS:
Behavioral: Cognitive-behavioral psychotherapy — The goal is to develop an internet and smart phone delivered CBT (iCBT) for the treatment of pediatric OCD on the bases of our feasibility study. This group will start directly with therapy of 16 weeks. The waiting group gets the same intervention after 16 weeks of waiting.

SUMMARY:
Internet-based psychotherapy for children and adolescents with obsessive-compulsive symptoms and an age of 6 to 18 years. Sessions are verified with teleconferencing with an psychotherapist, children and their parents. The psychotherapy is supported by an App and a wristband to obtain psychophysiological data. The investigators have already successfully performed a feasibility study.The goal of the current proposal is to develop an internet and smart phone delivered CBT (iCBT) for the treatment of pediatric OCD on the bases of the feasibility study. Internal testing on iCBT therapy package and developmental workchanges has been done. The investigators are now evaluating effectiveness in an RCT.

DETAILED DESCRIPTION:
In this study the investigators test effectiveness of an internet-based therapy approach for children with obsessive-compulsive disorders in an RCT design with a waiting control group. The investigators are planninng the investigation of 20 patients in each group.Therapy is verified by experts via teleconferences and a therapy app. Outcomes for the treatment group are evaluated before randomization (baseline, t0), 16 weeks (end of treatment, t1), 32 weeks (follow-up 1, t2), and 48 weeks after randomization (follow-up 2, t3). For the waiting list-group, outcomes are measured before the first randomization (baseline), at 16 weeks (waiting list period), 32 weeks (end of treatment), 48 weeks after the first randomization (follow-up I) and 64 weeks after the first randomization (follow-up II).

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents (ages 6-18) with a primary DSM-5 obsessive-compulsive disorder and at least 1 primary caretaker
* German-speaking (child & caretakers)
* Family home equipped with broadband connection and appropriate computer, monitor, HD webcam, and speaker and smart phone
* written informed content of the child and his caretaker
* OCD as highest treatment priority

Exclusion Criteria:

* IQ below 70
* not speaking and understanding German
* A psychiatric comorbidity that makes participation clinically inappropriate (for example, primary anorexia nervosa), depression with suicidality, psychosis or any other psychiatric disorder that requires acute treatment

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Schedule for Affective Disorders and Schizophrenia for School-Age Children Present and Lifetime Version (K-SADS-PL) | baseline,16 weeks, 32 weeks, 48 weeks, 64 weeks
  Clinical interview for psychiatric disorders for children and parents.
Change in Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) | baseline,16 weeks, 32 weeks, 48 weeks, 64 weeks
  Interview/questionnaire for obsessive-compusive disorders.
Change in Children's Global Assessment Scale (CGAS) | baseline,16 weeks, 32 weeks, 48 weeks, 64 weeks
  The CGAS is a measure of level of functioning in children and adolescents.
Change in Child Behavior Checklist (CBCL/6-18R) | baseline,16 weeks, 32 weeks, 48 weeks, 64 weeks
  A 113-item 3-point questionnaire for parents that assesses a wide range of child behavioral and emotional problems.
Change in Questionnaire for Measuring Health-Related Quality of Life in Children and Adolescents (KINDL) | baseline,16 weeks, 32 weeks, 48 weeks, 64 weeks
  A 24 item 5 point scale self-report questionnaire for children and parents to quality of life.
Change in Child Obsessive Compulsive Disorder Impact Scale (COIS-RC) | baseline,16 weeks, 32 weeks, 48 weeks, 64 weeks
  A 33-item self-report questionnaire to the impact of OCD symptoms on the psychosocial functioning of the children.
Change in Youth Self-Report (YSR/11-18R) | baseline,16 weeks, 32 weeks, 48 weeks, 64 weeks
  A 112 item 3-point scale completed by the children themselves and addresses a variety of behavioral and emotional problems.
Change in Depression Inventory for Children and Adolescents (DIKJ) | baseline,16 weeks, 32 weeks, 48 weeks, 64 weeks
  The questionnaire measures depressive symptoms in the children. It has 26 items and a 4 point scale.
Change in Junior temperament and character inventory (JTCI) | baseline,16 weeks, 32 weeks, 48 weeks, 64 weeks
  The questionnaire assesses temperament characteristics with 103/86 items and a 5-point scale.
Change in Screen for Child Anxiety Related Emotional Disorders (SCARED) | baseline,16 weeks, 32 weeks, 48 weeks, 64 weeks
  The SCARED assesses DSM-IV anxiety symptoms.
Change in Clinical Global Impressions-Severity (CGI-S) | baseline,16 weeks, 32 weeks, 48 weeks, 64 weeks
  A clinical 7-point rating scale of symptom severity.
Change in Clinical Global Impressions-Improvement (CGI-I) | baseline,16 weeks, 32 weeks, 48 weeks, 64 weeks
  A clinical 7-point rating scale of symptom severity.
Change in Impairment by OCD symptoms | Every day throughout the therapy process
  Children and parents indicate impairment by OCD via app.
Change in Extend of avoidance behavior | Every day throughout the therapy process
  Children and parents indicate extend of avoidance behavior via app.
Change in Daily mood | Every day throughout the therapy process
  Children indicate their mood via app.
Change in How the day has been | Every day throughout the therapy process
  Children indicate how good the day has been via app.
Change in How strong OCD is | Every day throughout the therapy process
  Children and parants indicate how strong OCD is via app.
Change in How the week has been | weekly throughout the therapy process
  Children and parants indicate how the week has been via app.
Change in Anxiety ratings during exposures | Every exposure throughout the therapy process
  Children indicate how high anxiety was during exposures via app.
Change in Heart rate variability | Every day throughout the therapy process
  Heart rate variability as an indicator of stress levels is assessed with wristbands.
Change in time the OCD takes | Every day throughout the therapy process
  Children and parants indicate how much time OCD takes via app.
Change in HEXACO- Personality Inventory-Revised (HEXACO-PI-R) | baseline,16 weeks, 32 weeks, 48 weeks, 64 weeks
  This questionnaire assesses the core personality traits of children.
Change in Engagement- Fragebogen | baseline,16 weeks, 32 weeks, 48 weeks, 64 weeks
  Questionnaire for emotional, cognitive and behavioral engagement at school with 5 items each.
Change in How convinced the patient of his/her OCD thoughts is | every exposure
  assessed by App
Change in Ulmer Life Quality Inventory for parents of chronically ill children(ULQIE) | baseline,16 weeks, 32 weeks, 48 weeks, 64 weeks
  Questionnaire to life quality of parents related to the impairment through the illness of the child.

OTHER OUTCOMES:
Trauma History Questionaire (THQ) | baseline
  This is a 5-point scale and 28 items that measures trauma experience such as sexual abuse or emotional neglect.
Essener Trauma Inventory for Children and Adolescents (ETI-KJ) | baseline
  This questionnaire measures posttraumatic symptoms.
Childhood trauma questionaire (CTQ) | baseline
  This is a 24-item measure to traumatic events.

CONTACTS AND LOCATIONS:
Overall Officials: Annette Conzelmann, Phd, Principal Investigator — Department of Child and Adolescent Psychiatry University of Tübingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Yes
We share study matterial and statistical outputs.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Any time before and after completion of the study for 10 years.
Access Criteria: Upon request.

REFERENCES:
- [Derived] Hollmann K, Hohnecker CS, Haigis A, Alt AK, Kuhnhausen J, Pascher A, Worz U, App R, Lautenbacher H, Renner TJ, Conzelmann A. Internet-based cognitive behavioral therapy in children and adolescents with obsessive-compulsive disorder: A randomized controlled trial. Front Psychiatry. 2022 Oct 18;13:989550. doi: 10.3389/fpsyt.2022.989550. eCollection 2022. PMID 36329915
- [Derived] Conzelmann A, Hollmann K, Haigis A, Lautenbacher H, Bizu V, App R, Nickola M, Wewetzer G, Wewetzer C, Ivarsson T, Skokauskas N, Wolters LH, Skarphedinsson G, Weidle B, de Haan E, Torp NC, Compton SN, Calvo R, Lera-Miguel S, Alt A, Hohnecker CS, Allgaier K, Renner TJ. Internet-based psychotherapy in children with obsessive-compulsive disorder (OCD): protocol of a randomized controlled trial. Trials. 2022 Feb 21;23(1):164. doi: 10.1186/s13063-022-06062-w. PMID 35189937